CLINICAL TRIAL: NCT03849989
Title: Expression of hSPCA1 and Ultrastructural Analysis of the Skin Before and After Laser Therapy in Hailey-Hailey Disease
Brief Title: M. Hailey-Hailey: hSPCA1 Expression and Skin Structure Upon Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 64815
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2019-02

CONDITIONS: Hailey Hailey Disease
MeSH Terms: conditions — Pemphigus, Benign Familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hailey-Hailey disease (Experimental): Patients with Hailey Hailey, diagnosis confirmed by histopathology or genetics, with therapy resistant skin lesions suitable for ablative lasertherapy.
  Skin biopsy specimens will be taken before and after lasertherapy at three time points.
  Before treatment:
  Affected skin 4 mm punch for immunofluorescence and RNA extraction 2 mm for electron microscopy Healthy skin within same anatomical region 4 mm punch for immunofluorescence and RNA extraction
  Immediately after treatment of the treated area:
  2 mm punch for histopathology
  Six weeks after treatment:
  Treated skin 4 mm punch for immunofluorescence and RNA extraction 2 mm for electron microscopy
  2mm punch biopsy of clinically uninvolved skin of the upper arm for electron microscopy
  Patients without Hailey-Hailey disease:
  2mm punch biopsy of skin of the upper arm for electron microscopy
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — Skin biopsy:
  Tissue samples will be taken by punch biopsy according to the daily routine of the Department of Dermatology of the Maastricht UMC+.
  Steps:
  * Skin desinfection with chlorhexidine digluconate 1% solution
  * Local anaesthesia with lidocaine hydrochloride 1%
  * Biopsy specimens are taken with sterile punch device (disposable biopsy punch delivered by kai medical)
  * Biopsy specimens are retrieved with sterile pincer and cut with sterile blade
  * Wound is stitched with a single transcutaneous stich using absorbable suture (vicryl 4.0).
  * Wound will be treated with R/ fusidic acid ointment 3 to 5 times per day for two weeks
  * In the first week after laser therapy the wound will be covered by R/ Urgotull non-adhesive gauze, R/ Cutisoft cotton non-sterile gauze and R/ Klinipress exsupad absorbing bandage.

SUMMARY:
Hailey-Hailey disease is a genetic acantholytic dermatosis characterized by continuous erosion of the skin that results in a burning, painful sensation and restricts the patient in daily life. This disorder results from a genetic defect in a calcium pump, i.e. the hSPCA1 pump. Calcium pumps are crucial for the processing of cell-cell adhesion proteins such as E-cadherin, part of desmosomes, the major glue between keratinocytes in skin epidermis. Today therapy is mainly focussed on symptom relief and prevention of secondary infection.

Ablative laser therapy is known to result in a speedy healing of the affected skin site within 2 weeks following laser therapy. The fact that the treated skin site remains clear from this acantholytic disorder in the months/years following ablation, regardless the existence of a germline mutation, suggests that an epigenetic modification occurs in the process of wound healing.

Objective: to (1) study the expression of hSPCA1 in keratinocytes before and after laser therapy and (2) verify the loss of acantholysis by immunohistochemistry and electron microscopy of cell-cell adhesions before and after laser therapy

ELIGIBILITY:
1.Inclusion criteria

1.1.Hailey-Hailey patients

Inclusion Criteria:

* Clinically diagnosed M. Hailey-Hailey as confirmed by histopathology and/or genetic analysis.
* Indication for ablative laser therapy
* >18 years old
* Informed consent

1.2. Patients without Hailey-Hailey disease

* >18 years old
* Clinically no symptoms of M. Hailey-Hailey
* Informed consent

Exclusion Criteria:

* <18 years old
* Treatment with tetracyclines, topical hormones or oral retinoids within the last 30 days preceding participation
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
hSPCA1 expression | Assessed at time point 0 weeks
  Expression of the hSPCA1 calcium pump in keratinocytes before ablative treatment
hSPCA1 expression | Assessed 6 weeks after ablative treatment
  Expression of the hSPCA1 calcium pump in keratinocytes after ablative treatment

SECONDARY OUTCOMES:
Ultrastructure of the skin before and after ablative treatment by electron microscopy and comparison to clinically uninvolved skin and skin of patients without Hailey-Hailey disease. | At 0 weeks and 6 weeks after ablative therapy
  Cell-to-cell adhesion and desmosome ultrastructure before and after ablative treatment by electron microscopy and comparison to clinically uninvolved skin and skin of patients without Hailey-Hailey disease.
Expression and localization of desmosomal proteins before and after ablative therapy by immunofluorescence. | At 0 weeks and 6 weeks after ablative therapy
  Expression and localization of desmosomal proteins before and after ablative therapy by immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Verstraeten, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hailey-Hailey disease and tight junctions: Claudins 1 and 4 are regulated by ATP2C1 gene encoding Ca(2+) /Mn(2+) ATPase SPCA1 in cultured keratinocytes. — https://www.ncbi.nlm.nih.gov/pubmed/22639968
- See also: Carbon dioxide laser treatment in Hailey-Hailey disease: a series of 8 patients. — https://www.ncbi.nlm.nih.gov/pubmed/23582735
- See also: The coexistence of Darier's disease and Hailey-Hailey disease symptoms. — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+coexistence+of+Darier's+disease+and+Hailey-Hailey+disease+symptoms.
- See also: Efficacy of erbium:YAG laser ablation in Darier disease and Hailey-Hailey disease. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Efficacy+of+erbium%3AYAG+laser+ablation+in+Darier+disease+and+Hailey-Hailey+disease
- See also: Carbon dioxide laser treatment for Hailey-Hailey disease: a retrospective chart review with patient-reported outcomes. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Carbon+dioxide+laser+treatment+for+Hailey-Hailey+disease%3A+a+retrospective+chart+review+with+patient-reported+outcomes.
- See also: Laser therapy for the treatment of Hailey-Hailey disease: a systematic review with focus on carbon dioxide laser resurfacing. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Laser+therapy+for+the+treatment+of+Hailey-Hailey+disease%3A+a+systematic+review+with+focus+on+carbon+dioxide+laser+resurfacing.